CLINICAL TRIAL: NCT05890313
Title: Pilot Study on Clinical Decision Support Tools for Referral for Dementia Consultation
Brief Title: Improving the Referral of Patients With Suspected Cognitive Impairment and Early Dementia
Acronym: DemRefImprov
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Unidade Local de Saúde de Matosinhos, EPE (Other); Instituto de Saude Publica da Universidade do Porto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DemRefImprov
Record Dates: First submitted 2023-05-15; First posted 2023-06-06 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-05

CONDITIONS: Cognitive Dysfunction; Mild Cognitive Impairment
Keywords: mild cognitive impairment; early dementia; timely diagnosis; primary care; referral process
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Intervention Model Description: The unit of study is the FHU. The six FHU recruited will be randomly allocated to the three study groups and each FHU will belong to the same group during the total period of the study. The study will be conducted simultaneously in all groups.
Who Masked: Care Provider
Masking Description: The pilot study is single blinded in the perspective of the Neurology consultation, regarding the origin and method of referral of each patient with a suspected diagnosis of MCI or early dementia from primary care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group MoCA/MMSE (Interventional Group) (Experimental): A training session about dementia management and standardized criteria for referral will be provided to participant PCCs, complemented with training in the administration of MMSE and MoCA, provided also to resident clinicians responsible for administration of the tests. MMSE will be administered if the patient has three to four years of schooling, and the MoCA will be used if the patient has more than four years of schooling. Patients with less than three years of education will be evaluated through regular clinical practice.
  Interventions: Diagnostic Test: Mini Mental State Examination; Diagnostic Test: Montreal Cognitive Assessment
- Group Brain on Track/MoCA/MMSE (Interventional Group) (Experimental): The training sessions mentioned in group MoCA/MMSE will be similarly provided in this group. Brain on Track is a web-based platform, used to remotely monitor cognitive function. There will be a first assessment with the aim of training eligible patients to correctly use Brain on Track, and a second assessment, one week after the first session. Depending on the score obtained in the second assessment, patients will be immediately referred to a specialized consultation, will not be referred or will be followed up during a period of 12 months with remote self monitorization, every three months. According to the total score from the four self-assessments performed in the follow-up period, PCCs will decide whether to refer or not. Patients who are illiterate will be evaluated through regular clinical practice, or MMSE or MoCA tests, according to years of schooling, if they are literate, but do not gather the inclusion criteria for the administration of Brain on Track.
  Interventions: Diagnostic Test: Mini Mental State Examination; Diagnostic Test: Montreal Cognitive Assessment; Device: Brain on Track (version BOT.0.0.0 03.03.2023)
- Control Group (No Intervention): Regular clinical practice complemented with the provision of standardized criteria for referring patients with a suspected diagnosis of MCI or early dementia to PCCs.

INTERVENTIONS:
Diagnostic Test: Mini Mental State Examination — MMSE is a clinically validated cognitive test, broadly used in healthcare and scientific settings, and it is administered to individuals with cognitive complaints suspected of cognitive decline whose educational literacy is of three to four years of schooling. It is validated in the general Portuguese population and can discriminate normal cognition from dementia.
  Other Names: MMSE
  Arms: Group Brain on Track/MoCA/MMSE (Interventional Group); Group MoCA/MMSE (Interventional Group)
Diagnostic Test: Montreal Cognitive Assessment — MoCA is a clinically validated cognitive test, broadly used in healthcare and scientific settings, and it is administered to individuals with cognitive complaints suspected of cognitive decline whose educational literacy is, at least, of four years of schooling. It is validated in general Portuguese population and can discriminate MCI from dementia.
  Other Names: MoCA
  Arms: Group Brain on Track/MoCA/MMSE (Interventional Group); Group MoCA/MMSE (Interventional Group)
Device: Brain on Track (version BOT.0.0.0 03.03.2023) — Brain on Track is a class I web-based software medical device, accessible on most platforms, including desktops and laptops. It is designed to allow periodic self-administered cognitive tests to be performed, enabling a cognitive assessment and continuous monitoring of the cognitive state of the patient remotely. It is based on the classic tests of neuropsychological assessment and allows assessing the main areas of cognition through a test lasting approximately 22 minutes. The stimuli that integrate each subtest are randomized between sessions, which reduces the effect of learning and allows the accomplishment of serial assessments.The test is available in three versions, adapted to different levels of schooling: 1-4 years, 5-9 years and 10+ years. The performance in each test is compared with normative population data and performance over time. For each test performed, Brain on Track presents a cumulative risk score for the presence of cognitive impairment.
  Other Names: BOT
  Arms: Group Brain on Track/MoCA/MMSE (Interventional Group)

SUMMARY:
The goal of this interventional study is to implement and evaluate the adhesion to two types of interventional strategies for assessing cognitive function, at Family Health Units (FHU), providing primary care clinicians (PCCs) with support to the decision process, regarding the referral of patients suspected of having mild cognitive impairment (MCI) or early dementia to the specialized consultation of Neurology at the public hospital services. The defined intervention strategies are the paper version of the cognitive tests MMSE and MoCA -group MoCA/MMSE -and the class I digital medical device web-based Brain on Track - group Brain on Track/MoCA/MMSE -, which will be compared with the regular clinical practice as the Control Group.

The main question it aims to answer is:

• the impact on the referral process of the implemented cognitive assessment strategies in the two interventional study groups compared with the Control Group.

Trained health professionals, at FHU, will administer the cognitive tests mentioned above to the eligible patients suspected of having MCI or early dementia, in the interventional groups and, according to the respective results and other criteria used during the consultation, PCCs will decide about the need of referral to the Neurology consultation. In the Control Group, health professionals will provide the regular clinical assistance practised in the respective FHU. If the referral occurs, the Neurology specialist will perform a complete clinical neuropsychological assessment of the referred patients and will validate the suspected diagnosis made at FHU.

Eligible patients with suspected MCI or early dementia will perform the cognitive tests according to the interventional study group, at the FHU or remotely. In the Control Group, eligible patients will be assisted through the daily clinical practice in the respective FHU.

The research team will compare the interventional study groups with the Control Group, to see if there is an improvement on the referral process in the interventional groups, compared with the Control Group .

DETAILED DESCRIPTION:
The pilot study has an exploratory quasi-experimental design. It is single blinded in the perspective of the Neurology consultation, regarding the origin and method of referral of each patient with a suspected diagnosis of MCI or early dementia from primary care.

The study will be implemented at six Portuguese FHU from Matosinhos. FHU will be similar in size, demographic composition, annual average of patients with cognitive complaints suspected of a diagnosis of MCI or early dementia, and annual average of referrals of patients with suspected MCI or early dementia to specialized care. FHU will be randomly allocated to the three study groups, existing two FHU in each group.

In each FHU, all PCCs will be invited to participate and all eligible patients will be proposed to be included in the study. The PCCs will assess the patient during a normal consultation and, whenever considered relevant, will decide to apply the referral strategy based on the support tools available. This will be a non-probabilistic consecutive sampling process of the general population, carried out by PCCs. An average of 20 to 30 patients are expected to be referred to the specialized care, after one year of recruitment, in each group.

The study groups are characterized as the following:

i) Group MoCA/MMSE: a training session about dementia management and standardized criteria for referral will be provided to the participant PCCs, complemented with training in the administration of MMSE and MoCA, provided also to resident clinicians responsible for administration of the tests. MMSE will be administered if the patient has three to four years of schooling, and the MoCA will be used if the patient has more than four years of schooling. Patients with less than three years of education will be evaluated through regular clinical practice.

ii) Group Brain on Track/MoCA/MMSE: a training session about dementia management and standardized criteria for referral will be provided to the participant PCCs, complemented with training in the administration of Brain on Track, MMSE, and MoCA, provided also to resident clinicians responsible for administration of the tests. Brain on Track is a class I digital medical device web-based, used to remotely monitor cognitive function: https://neuroinova.com/brain-on-track/. There will be a first assessment that will have the aim of providing training to patients by a resident clinician. One week later, a second assessment will be performed. Depending on the score obtained in the second session, patients will be immediately referred to a specialized consultation, will not be referred or will be followed up during a period of 12 months with remote self monitorization, every three months. Concerning the patients followed-up, according to the total score from the four self-assessments, PCCs will decide whether to refer or not. Patients who are illiterate will be evaluated through regular clinical practice, or MMSE or MoCA tests, according to years of schooling, if they are literate, but do not gather the inclusion criteria for the administration of Brain on Track.

iii) Control group: regular clinical practice complemented with the provision of standardized criteria for referring patients with a suspected diagnosis of MCI or early dementia to PCCs.

In each study group, the participating health professionals will receive adequate training from the research team.

All referred patients will undergo a comprehensive neuropsychological assessment and a complete etiological study, performed by Neurologists from the reference hospital associated with the participating FHU. This assessment will validate the PCCs´ clinical decision of referral as correct or incorrect, in all three groups. Concerning the validation of the clinical decision of non-referral, all the patients not referred will be contacted by phone, one year after the participation in the study, to check if the diagnosis changed during that period of time and the patient is being followed up or will start to be followed up by a Neurologist.

Additionally, Focus Groups will be performed at the end of the period of patients´ recruitment of one year, with health professionals from FHU allocated to interventional groups, and at the end of the one-year follow-up period with Brain on Track, with patients who were allocated to this follow-up. The aim of this qualitative study is to perceive the experience of health professionals and patients on using the respective interventional cognitive strategies.

The success of the implementation of the study will be quantified by quality indicators of two types, indicators of adhesion and indicators of referral, which will be constructed upon data collected by PCCs in specific forms designed by the research team and integrated into the local computer network of FHU, as well as data collected by Neurologists in specific forms also created by the research team.

The statistical analysis of will be performed using SPSS statistical software and will consist of a comparison of the primary endpoints between the three study groups, using an adequate statistical test for independent samples, namely a Qui-Square test or a T-test. The significance level will be fixed at 5%. Concerning the secondary endpoint related to the adhesion to the interventional strategies implemented, models of logistic regression will be used to assess the associations between patients and health professionals sociodemographic and professional characteristics, and the level of adhesion to the intervention. Odds ratio with 95% confidence intervals will be computed using logistic regression. The qualitative data obtained from Focus Groups will be analyzed using NVivo software and all the information collected will be transcribed verbatim, and a thematic analysis and data triangulation will be performed subsequently.

ELIGIBILITY:
Inclusion Criteria:

* Adults who are native from Portugal and fluent in Portuguese, have not already been diagnosed with dementia, have no motor, visual and/or hearing limitations and present to PCCs with cognitive complaints
* In group Brain on Track/MoCA/MMSE, related to Brain on Track: have a computer and/or tablet at home, with internet access, and have minimal computer literacy, in addition to the previous referred inclusion criteria

Exclusion Criteria:

* Motor, visual and hearing limitations

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Positive predictive value of the implemented interventional strategies | 18 months
  To determine the capacity of MMSE, MoCA and Brain on Track of detecting the true positive cases of MCI among the total positive cases of suspected cognitive impairment
Adhesion of PCCs to the three cognitive interventions implemented | 12 months
  Number of MoCA/MMSE/Brain on Track tests prescribed by PCCs to the recruited patients (with inclusion criteria and who accept to participate in the study) per month
Adhesion of patients to remote monitorization with Brain on Track | 12 months
  Number of remote monitorization sessions with Brain on Track accomplished by each patient allocated to the follow-up period of 12 months/4
Referrals decided by PCCs in all study groups | 24 months
  Number of referrals decided by PCCs in each study group of patients who are eligible and accept to participate in the study, per month
Average number of MoCA/MMSE/Brain on Track tests prescribed by PCCs in the 12-month period of implementation/Average number of MoCA/MMSE/Brain on Track tests prescribed by PCCs at baseline | 12 months
  Evaluation of the adhesion to the cognitive tests implemented during the 12-month period of the study in comparison to the adhesion existent before the implementation of the study
Average number of referrals decided by PCCs in each group of the study in the total temporal period of the study/Average number of referrals decided by PCCs at baseline | 24 months
  Evaluation of the impact of the implemented interventions on the quantity of referred patients suspected of a diagnosis of MCI or early dementia, during the 12-month period of implementation, taking into account the comparison to the same average quantity before the implementation of the study
Number of referrals decided by PCCs based mainly on the result of the cognitive intervention administered/Total number of decisions of referral * 100 | 24 months
  Evaluation of the impact of the result obtained from the cognitive interventions administered on the clinical decision of referral made by PCCs
Number of correct referrals decided by PCCs based mainly on the result of the cognitive intervention administered/Number of correct referrals decided by PCCs in the Control group * 100 | 36 months
  Evaluation of the impact of the cognitive interventions administered and their result on the clinical decision of referral made by PCCs in comparison to the impact of regular clinical practice on the same type of clinical decision
Proportion of new cases diagnosed with dementia, in the different stages of progression: mild, moderate and severe | 18 months
  To determine the proportion of incident cases of dementia, from early to severe stages, among the patients referred to specialized care

SECONDARY OUTCOMES:
Adhesion to interventional strategies by health professionals | At one-year of recruitment
  Description of the experiences from health professionals, concerning the application of interventions in interventional groups, through Focus Groups
Adhesion to Brain on Track by patients allocated to remote follow-up | At the end of the remote monitoring period of 12 months with Brain on Track
  Description of the experiences from patients allocated to self-monitoring with Brain on Track during one year, through Focus Groups

CONTACTS AND LOCATIONS:
Overall Officials: Luís Ruano, PhD, Principal Investigator — Institute of Public Health of University of Porto
Locations (1):
- Instituto de Saúde Pública da Universidade do Porto, Porto, Portugal